CLINICAL TRIAL: NCT02756065
Title: Connectomics in Psychiatric Classification
Brief Title: Connectomics in Psychiatric Classification of Bipolar Disorder and Schizophrenia
Status: Completed | Type: Observational
Sponsor: Washington University Early Recognition Center (Other)
Responsible Party: Sponsor
Other Study IDs: 201404123
Record Dates: First submitted 2015-06-17; First posted 2016-04-29 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: Bipolar; schizophrenia; schizoaffective
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Individuals between 18-30 years old No diagnosis of Bipolar Disorder or Schizophrenia No intervention used
  Interventions: Other: no intervention
- Bipolar Disorder: Individuals between 18-30 years old Diagnosis of Bipolar Disorder No intervention used
  Interventions: Other: no intervention
- Schizophrenia: Individuals between 18-30 years old Diagnosis of Schizophrenia or Schizoaffective Disorder No intervention used
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention is used

SUMMARY:
Washington University Early Recognition Center is conducting a research study to examine brain functional connectivity and network patterns in participants with bipolar disorder and schizophrenia.

DETAILED DESCRIPTION:
This study extends the assessment of brain connectivity and function, being conducted in the Human Connectome Project (HCP), to psychiatrically ill populations. The HCP consortium has made significant improvements in MRI instrumentation, data acquisition, preprocessing, and analysis. These improvements are currently providing publicly available data on the structure, function, and connectivity of young adult human (age 22-35) brains at unprecedented spatial resolution, temporal resolution, and accuracy. This study will focus on individuals aged 18-40 years who have a diagnosis of either schizophrenia/schizoaffective disorder or bipolar disorder, or are healthy controls. Additionally, similar to the HCP, the investigator will study the effect of genetics on the patterns of brain connectivity in various psychiatric populations. DNA will be collected non-invasively from saliva. Furthermore, this investigator will study cortisol levels in hair samples as an additional assessment to help characterize brain imagining findings.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-30

Exclusion Criteria:

* Head Injury
* Unstable Medical Condition

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals between the ages of 18-30 with a diagnosis of Bipolar Disorder or Schizophrenia
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2014-09; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
MRI Brain Imaging | within one month of study enrollment
  The current project aims to uncover latent, homogenous, connectivity phenotypes using neuroimaging tools, which are free from the limitations of traditional diagnostic boundaries, and which correlate with clinical characteristics. The investigator will use resting state functional connectivity MRI (rs-fcMRI), diffusion MRI (dMRI) and tract-based spatial statistics (TBSS) to identify brain signatures that cut across schizophrenia (SZ) and bipolar (BP).

SECONDARY OUTCOMES:
DNA testing through saliva | within one month of study enrollment
  Saliva samples will be collected from participants for DNA extraction and the development of lymphoblastoid cell lines. DNA is used for research purposes only, for studies assessing brain connectivity in schizophrenia, bipolar disorder and control subjects.
Hair sample for cortisol measurement | within one month of study enrollment
  To see how cortisol levels can help characterize brain imaging findings

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mamah, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No